CLINICAL TRIAL: NCT05390138
Title: A Smart Sleep Apnea Self-management Support Programme(4S) to Improve Apnea Severity and Cardiovascular Health - A Pragmatic Randomized Controlled Trial With Mixed-method Evaluation
Brief Title: A Smart Sleep Apnea Self-management Support Programme(4S) for Subjects With Sleep Apnea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Agnes Yuen-Kwan Lai, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UW 21-135
Record Dates: First submitted 2022-04-21; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: This is a 2-group randomisation controlled trial with 4-month and 12-month follow-up. The Experimental group will receive 4S intervention in relation to self-management and the Control group will receive general hygiene information.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor did not aware of which groups the patients belongs to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smart Sleep Apnea Self-management Support Programme (4S) (Experimental): Patients will receive Smart Sleep Apnea Self-management Support Programme (4S) in addition to usual care
  Interventions: Behavioral: Smart Sleep Apnea Self-management Support Programme (4S)
- General Hygiene Information (GH) (Placebo Comparator): Patients will receive general hygiene information (GH) in addition to usual care
  Interventions: Behavioral: General Hygiene Information (GH)

INTERVENTIONS:
Behavioral: Smart Sleep Apnea Self-management Support Programme (4S) — The experimental group will receive usual care and Smart Sleep Apnea Self-management Support Programme (4S). The 4S includes two interview sessions, instant messages, phone calls, continuous personalized chat-based messaging and phone call support and hotline services in relation to self-management. An e-platform will be used for self-monitoring and group sharing sessions will be conducted for experience sharing.
  Other Names: 4S group
  Arms: Smart Sleep Apnea Self-management Support Programme (4S)
Behavioral: General Hygiene Information (GH) — The control group will receive usual care and general hygiene information (GH). The GH includes two GH sessions, instant messages, phone calls, continuous personalized chat-based messaging and phone call support and hotline services in relation to general hygiene information. An e-platform will be used for self-monitoring and group sharing sessions will be conducted for experience sharing.
  Other Names: GH group
  Arms: General Hygiene Information (GH)

SUMMARY:
OSA is a chronic disease with high prevalence that parallels with increasing obesity. Self-management programmes are perceived to be cost-effective in long-term OSA patient care and can supplement regular medical treatments. The current study attempt to examine the effectiveness of 4S on improving apnea severity, cardiovascular health and quality of life in 4S intervention (4S) group, compared to the general hygiene (GH) control group.

DETAILED DESCRIPTION:
OSA is a chronic disease with high prevalence that parallels with increasing obesity. OSA affects around 12% and 24% of adults in Hong Kong and China Mainland, respectively. Chronic intermittent hypoxia and sleep fragmentation of OSA leads to cardiometabolic and neurocognitive sequelae (e.g. hypertension, diabetes, daytime sleepiness and depression). Long-term, multidisciplinary management involving patients in decision-making of treatment strategies, shifting from positive airway pressure (PAP) device-focused to the patient-centered chronic care model has been suggested.

Mobile instant messaging (such as WhatsApp/WeChat) are popular and inexpensive for interactive messaging. Smartphone-based self-management interventions were reported improved self-efficacy and clinical outcomes in patients with chronic diseases. The investigator only found one mobile health application to support CPAP therapy for OSA and one ongoing trial of OSA self-management telematic support to improve CPAP adherence. There is underutilization of mobile technology in patient-centered self-management programmes to improve PAP treatment and lifestyle modifications in OSA.

The current study attempt to examine the effectiveness of 4S on improving apnea severity, cardiovascular health and quality of life in 4S intervention (4S) group, compared to the general hygiene (GH) control group. Questionnaire and simple fitness assessment will be used to assess the effectivness of the intervention at 4-month and 12-month follow-up. Focus group interview will be conducted to collect qualiatative feedback on the intervention.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years and above;
* diagnosis of moderate to severe obstructive sleep apnea (AHI≥15);
* physically inactive (self-reported moderate physical activity per week of <150 minutes);
* overweight (BMI≥23 kg/m2);
* mentally, cognitively and physically fit to join the trial as determined by the doctor in-charge and responsible clinical investigators;
* able to speak and read Chinese;
* willing to complete the questionnaires and assessments;
* has a smartphone with instant messaging function (eg. WhatsApp/WeChat); and
* willing to give informed consent.

Exclusion Criteria:

* sleep disorder other than OSA;
* clinically significant psychiatric, neurological, or medical disorder other than OSA; and
* use of prescription drugs or clinically significant drugs affecting sleep.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2024-09-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Change in apnea hypopnea index | Baseline, 4 months
  Apnea hypopnea index will be asssessed by sleep test. The apnea hypopnea index is the number of times of apnea or hypopnea during one night, divided by the hours of sleep. The higher the apnea hypopnea index, the more severe sleep apnea is.

SECONDARY OUTCOMES:
Change in apnea hypopnea index | Baseline and 12 months
  Apnea hypopnea index will be assessed by sleep test. The apnea hypopnea index is the number of times of apnea or hypopnea during one night, divided by the hours of sleep. The higher the apnea hypopnea index, the more severe sleep apnea is.
Change in Duration of <90% oxygen desaturation | Baseline, 4 months and 12 months
  Duration of <90% oxygen desaturation will be assessed by sleep test.
Change in body weight | Baseline, 4 months and 12 months
  Body weight will be measured.
Change in body fat | Baseline, 4 months and 12 months
  Body fat will be measured.
Change in body neck circumference | Baseline, 4 months and 12 months
  Neck circumference will be measured.
Change in waist circumference | Baseline, 4 months and 12 months
  Waist circumference will be measured.
Change in hip circumference | Baseline, 4 months and 12 months
  Hip circumference will be measured.
Change objective physical activity level | Baseline, 4 months and 12 months
  Steps count and acceleration pattern of physical activity will be measured by a 7-day waist-worn accelerometer.
Change in Hand grip strength | Baseline, 4 months and 12 months
  Hand grip strength will be measured by a dynamometer.
Change in lower limb strength | Baseline, 4 months and 12 months
  Lower limb strength will be measured by a 30-second chair stand test.
Change in flexibility | Baseline, 4 months and 12 months
  Flexibility will be measured by a sit and reach test.
Change in balance | Baseline, 4 months and 12 months
  Balance will be measured by a single-leg stance test.
Change in daytime sleepiness | Baseline, 4 months and 12 months
  Daytime sleepiness will be measured by a 8-item Epworth Sleepiness Scale with a 3-point Likert scale. Total scores range from 0 to 24. Higher scores reflect greater daytime sleepiness.
Change in sleep quality | Baseline, 4 months and 12 months
  Sleep quality will be measured by a 7-item Insomnia Severity Index with a 4-point Likert scale. Total scores range from 0 to 28. Higher scores reflect greater severity of insomnia.
Change in functional outcomes of sleep | Baseline, 4 months and 12 months
  Functional outcomes of sleep will be measured by 10-item Functional Outcomes of Sleep Questionnaire with a 4-point Likert scale. Total scores range from 10 to 40. Higher scores reflect better functional outcomes of sleep.
Change in quality of life | Baseline, 4 months and 12 months
  Quality of life will be measured by 5-item EuroQol 5-Dimension questionnaire. The EQ-5D descriptive system is a preference-based HRQL measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Change in anxiety symptoms | Baseline, 4 months and 12 months
  Anxiety symptoms will be measured by Generalised Anxiety Disorder Assessment (GAD-7) with a 3-point Likert scale. Total scores range from 0 to 21. Higher scores reflect more higher anxiety symptoms.
Change in depressive symptoms | Baseline, 4 months and 12 months
  Depressive symptoms will be measured by 9-item Patient Health Questionnaire-9 (PHQ-9) with a 3-point Likert scale. Total scores range from 0 to 27. Higher scores reflect more higher depressive symptoms.
Change in subjective happiness | Baseline, 4 months and 12 months
  Subjective happiness will be measured by 4-item Subjective Happiness Scale with a 7-point Likert scale. Total scores range from 4 to 28. The highest scores reflect greater happiness.
Change in subjective physical activity level | Baseline, 4 months and 12 months
  Subjective physical activity level will be measured by 8-item International Physical Assessment Questionnaire -short version
Change in dietary habits | Baseline, 4 months and 12 months
  Dietary habits will be measured by 10-item dietary intake and practice questionnaire.
Change in self-efficacy in CPAP use | Baseline, 4 months and 12 months
  Self-efficacy in CPAP use will be measured by a 26-item Self-efficacy Measure for Sleep Apnea. Each Item ranges from 1 to 4: Higher scores indicate greater perceived self-efficacy, greater perceived response efficacy, and higher perceived susceptibility.
Change in exercise and dietary control self-efficacy | Baseline, 4 months and 12 months
  Exercise and dietary control self-efficacy will be measured by outcome-based questionnaire. Each item ranges from 1-10. The higher scores indicate higher self-efficacy
Change in perceived support from family and peers | Baseline, 4 months and 12 months
  Perceived support from family and peers measured by a 8-item Multidimensional Scale of Perceived Social Support with a 7-point Likert scale. Total scores for both family and peer subscales range from 4 to 28. Higher scores reflect better perceived social support.
Change in patient activation | Baseline, 4 months and 12 months
  Knowledge, skills and confidence in self-management were measured by a 13-item Patient Activation Measure Scale. The total score ranges from 0 (no activation) to 100 (high activation), with higher scores denoting the better patient activation.
Intervention credibility | 4 months and 12 months
  The rationale of the delivered treatment and its efﬁcacy to alleviate sleep apnea will be measured using the 4-item Credibility of Treatment Rating Scale. Each item ranges from 1-6. The higher scores indicate higher credibility.

CONTACTS AND LOCATIONS:
Overall Officials: Agnes YK Lai, PhD, Principal Investigator — The University of Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Need to obtain consent from patients before agreeing to share individual participants data.
Supporting Information: Study Protocol
Time Frame: When study finished
Access Criteria: The minimal anonymized dataset will be available upon request to interested researchers. For interested researchers, please contact, Mr George Cheung (email ocgeorge@hku.hk), (School of Nursing, The University of Hong Kong) for further information.

REFERENCES:
- [Background] Benjafield AV, Ayas NT, Eastwood PR, Heinzer R, Ip MSM, Morrell MJ, Nunez CM, Patel SR, Penzel T, Pepin JL, Peppard PE, Sinha S, Tufik S, Valentine K, Malhotra A. Estimation of the global prevalence and burden of obstructive sleep apnoea: a literature-based analysis. Lancet Respir Med. 2019 Aug;7(8):687-698. doi: 10.1016/S2213-2600(19)30198-5. Epub 2019 Jul 9. PMID 31300334
- [Background] Epstein LJ, Kristo D, Strollo PJ Jr, Friedman N, Malhotra A, Patil SP, Ramar K, Rogers R, Schwab RJ, Weaver EM, Weinstein MD; Adult Obstructive Sleep Apnea Task Force of the American Academy of Sleep Medicine. Clinical guideline for the evaluation, management and long-term care of obstructive sleep apnea in adults. J Clin Sleep Med. 2009 Jun 15;5(3):263-76. PMID 19960649
- [Background] Andrade FM, Pedrosa RP. The role of physical exercise in obstructive sleep apnea. J Bras Pneumol. 2016 Nov-Dec;42(6):457-464. doi: 10.1590/S1806-37562016000000156. PMID 28117479
- [Background] Iftikhar IH, Kline CE, Youngstedt SD. Effects of exercise training on sleep apnea: a meta-analysis. Lung. 2014 Feb;192(1):175-84. doi: 10.1007/s00408-013-9511-3. PMID 24077936
- [Background] Aiello KD, Caughey WG, Nelluri B, Sharma A, Mookadam F, Mookadam M. Effect of exercise training on sleep apnea: A systematic review and meta-analysis. Respir Med. 2016 Jul;116:85-92. doi: 10.1016/j.rmed.2016.05.015. Epub 2016 May 21. PMID 27296826
- [Background] Stepnowsky CJ, Palau JJ, Gifford AL, Ancoli-Israel S. A self-management approach to improving continuous positive airway pressure adherence and outcomes. Behav Sleep Med. 2007;5(2):131-46. doi: 10.1080/15402000701190622. PMID 17441783
- [Background] Dickerson SS, Jungquist C, TenBrock E, Aquilina A, Smith P, Sabbah EA, Alameri R, Dean G. Feasibility Testing of a Self-Management Program Book to Improve Adherence to PAP in Persons Newly Diagnosed With Sleep Apnea. Behav Sleep Med. 2018 Sep-Oct;16(5):413-426. doi: 10.1080/15402002.2016.1228644. Epub 2016 Sep 23. PMID 27660897
- [Background] Dickerson SS, TenBrock E, Smith P, Kwon M, Chacko T, Li CS, Dean GE. Mixed methods feasibility study of Breathe2Sleep a peer modeling approach to PAP self-management. Heart Lung. 2020 Nov-Dec;49(6):949-958. doi: 10.1016/j.hrtlng.2020.04.015. Epub 2020 May 28. No abstract available. PMID 32473747
- [Background] Zimbudzi E, Lo C, Misso ML, Ranasinha S, Kerr PG, Teede HJ, Zoungas S. Effectiveness of self-management support interventions for people with comorbid diabetes and chronic kidney disease: a systematic review and meta-analysis. Syst Rev. 2018 Jun 13;7(1):84. doi: 10.1186/s13643-018-0748-z. PMID 29898785
- [Background] Suarez-Giron M, Garmendia O, Lugo V, Ruiz C, Salord N, Alsina X, Farre R, Montserrat JM, Torres M. Mobile health application to support CPAP therapy in obstructive sleep apnoea: design, feasibility and perspectives. ERJ Open Res. 2020 Feb 10;6(1):00220-2019. doi: 10.1183/23120541.00220-2019. eCollection 2020 Jan. PMID 32055630